CLINICAL TRIAL: NCT04202419
Title: Clinical Evaluation of a Nonablative Fractional 1940 nm Diode Laser for Treatment of Pigmented Lesions
Brief Title: Nonablative Fractional Diode Laser for Treatment of Pigmented Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Collaborators: Miami Dermatology and Laser Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRX19005
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Pigmented Skin Lesion
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Group (Experimental): Single Arm: All subjects will undergo treatment of pigmented lesions with a 1940 nm diode laser
  Interventions: Device: FRAX 1940 nm laser

INTERVENTIONS:
Device: FRAX 1940 nm laser — A fractional 1940 nm solid-state diode laser will deliver linear arrays of microbeams to create nonablative microscopic treatment zones (MTZs) in the skin, in order to treat pigmented skin lesions.

SUMMARY:
This study is being conducted to evaluate the safety and efficacy of a fractional diode laser for treatment of pigmented lesions such as, but not limited to lentigos (age spots), solar lentigos (sunspots), and ephelides (freckles).

DETAILED DESCRIPTION:
Prospective, open-label, clinical trial to study the effects of the nonablative, fractional diode laser for treatment of pigmented lesions.

Up to 60 eligible participants will be enrolled at up to five (5) sites. Participants will receive up to three (3) treatments in the following treatment areas: face, hands, arms, back, chest, or legs. Participants will complete follow-up visits for clinical evaluation and photography at 1 and 3 months after the final study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 21 to 70
3. Fitzpatrick Skin Type I to VI
4. Willingness to have test spots and up to three (3) treatments for pigmented lesions on or off the face which are rated at baseline as moderate or higher per Investigator or study staff
5. Provide signed informed consent to participate in the study
6. Adhere to study treatment and follow-up schedules
7. Willing to have hair removed from the intended treatment area prior to treatment and/or photography
8. Avoid sun exposure to all treated areas and use of sunscreen with sun protection factor (SPF) 30 or greater throughout the duration of the study
9. Adhere to post-treatment care instructions
10. Allow photography of treated areas and to release their use for scientific and/or promotional purposes

Exclusion Criteria:

1. Pregnant, planning to become pregnant, or breast feeding during the study
2. Allergy to lidocaine or similar medications
3. Excessively tanned skin in the intended treatment area
4. Open wound or infection in the intended treatment area
5. Tattoo(s) or permanent make-up in the intended treatment area
6. Skin condition in the intended treatment area that could interfere with treatment or evaluation of safety or efficacy
7. Presence or history of melasma
8. Presence or history of skin cancer within the treatment area
9. History of keloid or hypertrophic scar formation
10. History of herpes simplex virus (HSV) or similar condition in the intended treatment area unless treated with prophylactic medication
11. Diagnosed coagulation disorder
12. Immunosuppression disorder
13. Presence of any medical condition that in the opinion of the Investigator could impair healing or outcome as a result of treatment
14. Use of systemic retinoid therapy (e.g. Accutane) during the past six (6) months
15. Use of topical retinoid therapy in the intended treatment area during the past two (2) weeks
16. Use of oral corticosteroid therapy during the past four (4) weeks
17. Prior treatment, such as surgery, light, laser or radiofrequency (RF) procedures in the intended treatment area during the past three (3) months
18. Prior injectable dermal fillers (e.g. collagen, hyaluronic acid) in the intended treatment area within the past 12 months
19. Prior injectable toxins (e.g. Botox) in the intended treatment area within the past three (3) months
20. Subjects who in the opinion of the Investigator are unwilling or unable to adhere to the study requirements, or who are otherwise not a good candidate for the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Waibel, M.D, Principal Investigator — Miami Dermatology and Laser Institute
Locations (1):
- Miami Dermatology and Laser Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nonablative Fractional Diode Laser: Single Arm: All subjects will undergo treatment of pigmented lesions with a 1940 nm diode laser
  FRAX 1940 nm laser: A fractional 1940 nm solid-state diode laser will deliver linear arrays of microbeams to create nonablative microscopic treatment zones (MTZs) in the skin, in order to treat pigmented skin lesions.
Period: Overall Study
Arm/Group | Nonablative Fractional Diode Laser
Started | 30
Completed | 20
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: Thirty subjects with 30 areas were enrolled in study FRX19005
Units Other Than Participants: treatment areas
Arm/Group | Single Group
Number analyzed (Participants) | 30
Number analyzed (treatment areas) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Pigmented Lesion Improvement by Blinded Evaluation
Description: The primary efficacy endpoint was defined as improvement in the clearance of pigmented lesions, as assessed by three (3) blinded evaluators comparing photographs taken at Baseline/Pre-treatment and at the 1-month follow-up (post final treatment)
Time Frame: 1 month follow-up post treatment series, where treatment could last up to 10 weeks after baseline
Population: Data from FRX19005 study was combined with FRX19004 study (NCT04203745) for ad-hoc primary efficacy analysis via blinded evaluation. Both trials assessed the 'treatment of pigmented lesions' and are directly comparable due to equivalence of patient populations and efficacy endpoints, therefore, the exact same analyses were performed. The treated area was considered a "success" if at least 2 of the 3 reviewers correctly identified the post-treatment photograph (i.e. left or right side).
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Nonablative Fractional Diode Laser
Number analyzed (Participants) | 56
Number analyzed (Observations) | 45
Observations | 41

2. Secondary Outcome: Pigmentation Improvement at the 3-month Follow-up, by Blinded Evaluation
Description: The secondary endpoint was pigmentation improvement at the 3-month follow-up, as assessed by three (3) blinded evaluators comparing photographs taken at Baseline/Pre-treatment and at the 3-month follow-up (post final treatment). The treated area was considered a "success" if at least two of the three reviewers correctly identified the post-treatment photograph (i.e. left or right side).
Time Frame: 3-months post final treatment, where treatment series could last up to 10 weeks after baseline
Population: Data from FRX19004 study was combined with FRX19005 study (NCT04202419) for ad-hoc primary efficacy analysis via blinded evaluation. 42 slides containing 1 pair of photos (taken pre-treatment and 3-months post-treatment) were presented to three blinded evaluators. The treated area was considered a "success" if at least 2 of the 3 reviewers correctly identified the post-treatment photograph (i.e. left or right side).
Measure: Count of Units; unit: observations
Units Other Than Participants: observations
Arm/Group | Nonablative Fractional Diode Laser
Number analyzed (Participants) | 56
Number analyzed (observations) | 42
observations | 35

3. Secondary Outcome: Blinded Assessment of Textural Improvement Using a 5-point Global Aesthetic Improvement Scale (GAIS)
Description: For each reviewer assessment: If the post-treatment photograph was identified correctly, the reviewer's assessment on the textural scale was coded as follows: -1=worse, 0=no change; 1=improved; 2=much improved; and 3=very much improved. If not identified correctly, the scale was reversed (-1=improved, 0=no change, 1=worsened, 2=much worsened and 3=very much worsened). Results were based on the majority rule of the assessments by the three blinded reviewers; in other words, the mode of the three blinded reviewers' scores was used as the treated area clearance results, while the median was used if three different scores were reported.
Time Frame: 1 month follow-up post treatment series, where treatment could last up to 10 weeks after baseline
Population: Data from FRX19005 study was combined with FRX19004 study (NCT04203745) for ad-hoc efficacy analysis via blinded evaluation. Both trials assessed the 'treatment of pigmented lesions' and are directly comparable due to equivalence of patient populations and efficacy endpoints, therefore, the exact same analyses were performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Nonablative Fractional Diode Laser
Number analyzed (Participants) | 45
Participants
  Worse | 1
  No change (stable) | 16
  Improved | 28

4. Secondary Outcome: Subject Assessment of Improvement Using a 5-point Global, Aesthetic Improvement Scale (GAIS)
Description: Subject assessments of treatment outcome were completed at the 1-month follow-up using the Global Assessment Improvement Scale (GAIS). The scale was coded as follows: -1=worse, 0=no change; 1=improved; 2=much improved; and 3=very much improved
Time Frame: 1 month follow-up post treatment series, where treatment could last up to 10 weeks after baseline
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nonablative Fractional Diode Laser
Number analyzed (Participants) | 45
Participants
  Worse | 1
  No Change | 3
  Improved | 17
  Much Improved | 10
  Very Much Improved | 14

5. Secondary Outcome: Subject Satisfaction With Treatment Results
Description: Subject satisfaction with treatment results completed at the 1-month follow-up using a 5 point scale coded as follows: -1=not satisfied, 0=little satisfied; 1=somewhat satisfied; 2=satisfied; and 3=very satisfied
Time Frame: 1 month follow-up post treatment series, where treatment could last up to 10 weeks after baseline
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nonablative Fractional Diode Laser
Number analyzed (Participants) | 44
Participants
  Not Satisfied | 1
  Little Satisfied | 2
  Somewhat Satisfied | 14
  Satisfied | 12
  Very Satisfied | 15

ADVERSE EVENTS:
Time Frame: 12 weeks following last treatment, where treatment series could last up to 10 weeks.
Arm/Group | Nonablative Fractional Diode Laser
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04202419/Prot_SAP_001.pdf